CLINICAL TRIAL: NCT03858712
Title: Nonrandomized Phase II Hybrid Type 3 Implementation Study: Feasibility and Acceptance of an EHR-embedded Oral Cancer Directed Therapy Toxicity and Adherence Program for Patients With Breast or Gastrointestinal Cancer
Brief Title: EHR-embedded OCDT in Breast or GI Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nadine McCleary MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-571
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Oral Cancer Directed Therapy; Breast Cancer; Gastrointestinal Cancer; Oral Chemotherapy
Keywords: Oral Cancer Directed Therapy; Breast Cancer; Gastrointestinal Cancer; oral chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: Hybrid type 3 implementation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive Care Team Alert (Other): DFCI patients with advanced breast or gastrointestinal cancer prescribed Oral Cancer Directed Therapy.
  * Screening: ePRO Clinic:-- complete ePRO clinic for all medical oncology scheduled provider appointments during the study period per standard practice
  * ePRO Home: -- ePRO oral between visits at home.
  * Passive care team alert -- EHR inBasket notification
  Interventions: Other: Passive Care Team Alert
- Active Care Team Alert (Other): DFCI patients with advanced breast or gastrointestinal cancer prescribed Oral Cancer Directed Therapy.
  * Screening: ePRO Clinic:-- complete ePRO clinic for all medical oncology scheduled provider appointments during the study period per standard practice
  * ePRO Home: -- ePRO oral between visits at home.
  * Active care team alert -- practice nurse monitoring of ePRO home responses score = 3 indicating a moderate-severe toxicity (grade 3 or higher
  Interventions: Other: Active Care Team Alert

INTERVENTIONS:
Other: Active Care Team Alert — 2) Active care team alert via office practice nurse monitoring of ePRO oral responses scored at 3, indicating moderate-severe (grade ≥3) toxicity.
  Office practice nurses will monitor ePRO oral responses and respond to those scored at 3 per disease center symptom management protocol.
  The ePRO oral responses from the remaining participants will additionally be monitored by office practice nurses who will respond to ePRO responses with scores of 3, indicating a moderate-severe toxicity (grade 3 or higher).
  Arms: Active Care Team Alert
Other: Passive Care Team Alert — Primary care teams are assigned an EHR inBasket pool through which PP messages are delivered. Providers will be responsible for reviewing ePRO responses via inBasket, selecting "mark as reviewed" button as mandated for all clinical messages within 48 hours per policy.
  Arms: Passive Care Team Alert

SUMMARY:
This is research study is for participants with advanced breast or gastrointestinal cancer who have been taking oral chemotherapy medication (Oral Cancer Directed Therapy). This study is to help researchers better understand gaps in assessing oral chemotherapy patient toxicity at home, adherence to treatment and integrate toxicity/adherence reporting.

DETAILED DESCRIPTION:
For patients with advanced breast or gastrointestinal cancer prescribed Oral Cancer Directed Therapy.

* Participants will complete ePRO clinic for all medical oncology scheduled provider appointments during the study period per standard practice
* Participants between clinic visits, will be asked to complete the oral weekly survey at home via the mobile or web based patient portal. The survey can be completed on a computer, tablet or smartphone at home or on a tablet at the time of scheduled visit.

  * The first 100 participants to complete the survey will receive a passive care team alert for responses (per DFHCC policy)
  * The second 100 participants to complete the survey will receive an active care team alert for responses.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 18 or older
* Male or Female
* Scheduled visit at DF/HCC within the BOC or GCC
* Diagnosis of advanced breast cancer or gastrointestinal cancer
* Prescribed any OCDT within prior 5 days of screening
* English as the primary language (as documented in the EHR, written or spoken, and patient interpreter needed flag = no)
* Mobile number listed in EHR to allow participation in ePP portion of the study
* Women of any pregnancy status
* Patients diagnosed with an advanced cancer will be eligible to participate in the study until discontinuation of OCDT or death, whichever occurs first

Exclusion Criteria

* Adults unable to provide verbal consent
* Pediatric patients
* Patients without access to a electronic device (including tablet, computer, aptop or smartphone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
ePRO Oral Response Rate | 30 days
  proportion of participants responding to at least 50% of ePRO oral questionnaires at 30 days

SECONDARY OUTCOMES:
ePRO Oral Response Rate | 60 days
  proportion of participants responding to at least 50% of ePRO oral questionnaires at 60 days
ePRO Oral Response Rate | 90 days
  proportion of participants responding to at least 50% of ePRO oral questionnaires at 90 days
Average number of ePRO oral questionnaires completed per week | 90 Days
  average number of ePRO oral questionnaires completed per week until discontinuation of OCDT or end of study (whichever occurs first)
Proportion of Participants reporting ePRO grade 3+ toxicity | 90 Days
  proportion of participants reporting grade 3+ toxicity on at least one ePRO oral questionnaire among participants who responded to at least one ePRO oral questionnaire
Proportion of Participants with an ePRO Intervention | 90 Days
  proportion of participants who were called by an office practice nurse for toxicity, had an OCDT dose modification, urgent clinic visit, ED visit or unplanned hospitalization among participants who responded to at least one ePRO oral questionnaire
Participant Report of OCDT Frequency | 90 Days
  proportion of participants who reported missing >20% of prescribed OCDT doses for reasons other than toxicity on at least one ePRO oral report among participants who responded to at least one ePRO oral questionnaire; measured by participant weekly report of dates and time (AM, PM) of missed doses of the prescribed OCDT regimen
Participant Report of OCDT Frequency | 30 Days
  Among participant who self-reported missing ≥20%/<20% of prescribed OCDT doses via ePRO oral, the proportion for whom EHR prescriptions also indicated non-adherence/adherence; EHR prescriptions measured by Proportion of Days Covered (PDC) = proportion of days covered by OCDT prescription claims divided by 30 days
ePRO oral willingness | 90 Days
  proportion of participants reporting that they were willing or very willing to use ePRO oral again in the future among participants who responded to at least one ePRO oral questionnaire
ePRO oral ease of use | 90 Days
  Proportion of participants reporting that ePRO oral was either easy or very easy to use among participants who responded to at least one ePRO oral questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nadine McCleary, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: http://www.dfhcc.harvard.edu/crs-resources/ODQ_Documents/02_CT.GOV_CTRP/Guidance_on_Data_Sharing.pdf